CLINICAL TRIAL: NCT02701153
Title: Phase II Study of 5-Day Hypofractionated Preoperative Radiation Therapy for Soft Tissue Sarcomas: Expansion Cohort
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Radiological Society of North America (Other); Sarcoma Alliance for Research through Collaboration (Other); Sarcoma Foundation of America (Unknown); Tower Cancer Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-001657; NCI-2016-00202 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-001657 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2016-03-02; First posted 2016-03-08 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Recurrent Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (hypofractionated radiation therapy) (Experimental): Patients undergo hypofractionated radiation therapy on Monday-Friday for 5 days. Beginning 2-12 weeks after completion of radiation therapy, patients undergo surgery.
  Interventions: Procedure: Conventional Surgery; Radiation: Hypofractionated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Conventional Surgery — Undergo surgery
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated Radiotherapy; hypofractionation
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the side effects of hypofractionated radiation therapy in treating patients with soft tissue sarcomas prior to surgery. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects.

DETAILED DESCRIPTION:
PRIMARY OBJCETIVES:

I. Grade >= 2 radiation morbidity (subcutaneous tissue fibrosis, joint stiffness, or edema) at 2 years.

SECONDARY OBJECTIVES:

I. Evaluate local control, regional control, distant metastasis, progression free survival, and overall survival.

II. Evaluate the functional outcomes as assessed using the musculoskeletal tumor rating scale (MSTS) and the Toronto Extremity Salvage Score (TESS).

III. Collect germ-line deoxyribonucleic acid (DNA) and nucleic acids from cancer patients to further investigate the association and identify new germ-line mutations that impact cancer predisposition.

IV. Investigate the role of germ-line mutations in predicting cancer outcome and response to therapy.

OUTLINE:

Patients undergo hypofractionated radiation therapy on Monday-Friday for 5 days. Beginning 2-12 weeks after completion of radiation therapy, patients undergo surgery.

After completion of study treatment, patients are followed up at 3 months and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed soft tissue sarcoma of the extremity/trunk
* Intermediate or high grade sarcoma
* Resectable primary lesion (patients with pre-existing metastasis will be included if their primary is still going to be resected)
* Recurrent, any grade, no previous radiation therapy
* Karnofsky performance status (KPS) >= 70 or Eastern Cooperative Oncology Group (ECOG) 0 - 2
* If a woman is of childbearing potential, a negative serum pregnancy test must be documented

Exclusion Criteria:

* Active treatment of a separate malignancy
* History of prior irradiation to the area to be treated
* Pre-operative chemotherapy (post-op acceptable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2016-02-03 (Actual); Primary Completion 2026-02-03 (Estimated); Study Completion 2027-02-03 (Estimated)

PRIMARY OUTCOMES:
Grade >= 2 radiation morbidity (subcutaneous tissue fibrosis, joint stiffness, or edema) | Up to 2 years
  Interim reports will be prepared every six months until the results of the study are published. In general, the interim reports will contain information about patient accrual rate with projected completion dates, status of question-answer (QA) review and compliance rate of treatment per protocol, and the frequencies and severity of toxicity.

SECONDARY OUTCOMES:
Distant metastasis | Up to 3 years
  Cumulative incidence approach (K-M plots and Cox proportional hazard modeling) will be used.
Local failure | Up to 3 years
  Cumulative incidence approach (Kaplan-Meier [K-M] plots and Cox proportional hazard modeling) will be used.
Overall survival | Up to 3 years
  Cumulative incidence approach (K-M plots and Cox proportional hazard modeling) will be used.
Progression free survival | Up to 3 years
  Cumulative incidence approach (K-M plots and Cox proportional hazard modeling) will be used.
Regional failure | Up to 3 years
  Cumulative incidence approach (K-M plots and Cox proportional hazard modeling) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Anusa Kalbasi, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Nikitas J, Kendal JK, Savjani RR, Jackson N, Peterson N, Deng J, Hernandez J, Chong N, Singh AS, Chmielowski B, Federman NC, Crompton JG, Kadera BE, Wessel LE, Christ AB, Nelson SD, Dry SM, Weidhaas JB, Steinberg ML, Bernthal NM, Eilber FC, Kalbasi A, Reddy VK. Five-Day Preoperative Radiation Therapy for Patients With High-Risk Soft Tissue Sarcoma: A Nonrandomized Clinical Trial. JAMA Netw Open. 2025 Dec 1;8(12):e2550195. doi: 10.1001/jamanetworkopen.2025.50195. PMID 41405883